CLINICAL TRIAL: NCT02336425
Title: A Multi-Center, Randomized, Double-Blind, Placebo- Controlled Study to Investigate the Efficacy and Safety of 52 Weeks Treatment With QGE031 Subcutaneous (s.c). in Asthma Patients Not Adequately Controlled by Medium- or High-dose Inhaled Corticosteroid (ICS) Plus Long Acting β2-agonist (LABA) With or Without Oral Corticosteroid (OCS)
Brief Title: Efficacy and Safety of QGE031 Compared With Placebo in Patients Aged 18-75 Years With Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to the efficacy results from an interim analysis (at the end of treatment epoch) of the Phase II study CQGE031B2201 (NCT01716754).
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQGE031B2204; 2014-003155-57 (EudraCT Number)
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — ligelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- QGE031 240 mg (Experimental): QGE031 240 mg subcutaneous injection every 4 weeks
  Interventions: Drug: QGE031
- QGE031 72 mg (Experimental): QGE031 72 mg subcutaneous injection every 4 weeks
  Interventions: Drug: QGE031
- QGE031 24 mg (Experimental): QGE031 24 mg subcutaneous injection every 4 weeks
  Interventions: Drug: QGE031
- Placebo to QGE031 (Placebo Comparator): Placebo subcutaneous injection every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QGE031 — QGE031 120 mg per 1 mL liquid in vial
  Arms: QGE031 24 mg; QGE031 240 mg; QGE031 72 mg
Drug: Placebo — Placebo to QGE031 0 mg per 1 mL liquid in vial
  Arms: Placebo to QGE031

SUMMARY:
This study planned to assess the effect on the reduction in rate of severe asthma exacerbations of different dose levels of QGE031 in asthma patients that are inadequately controlled with inhaled steroid plus beta-2 agonist medication with or without oral steroid. However, this study was terminated due to the efficacy results from an interim analysis (at the end of treatment epoch) of the Phase II study CQGE031B2201 (NCT01716754). Planned data analyses were not performed for this study due to the early termination and the very limited dataset (only 10 participants received study medication of the 440 participants planned).

ELIGIBILITY:
Key Inclusion Criteria:

* A diagnosis of allergic asthma, uncontrolled on current medication.
* History of at least 2 asthma exacerbations during the last 1 year
* Forced Expiratory Volume in one second (FEV1) of ≥ 40% and ≤ 80% of the predicted normal value; reversibility following administration of bronchodilator.

Key Exclusion Criteria:

* Use of tobacco products within the previous 6 months (Social occasional smokers may be included).
* Recent asthma attack/exacerbation or asthma worsening/ respiratory infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (3):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Kingwood, Texas
  - Novartis Investigative Site, Plano, Texas
- Novartis Investigative Site, Erpent, Belgium
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Novartis Investigative Site, Le Kremlin-Bicêtre, France
- Germany (7):
  - Novartis Investigative Site, Cottbus, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Münster
- Hungary (2):
  - Novartis Investigative Site, Miskolc, HUN
  - Novartis Investigative Site, Balassagyarmat
- Novartis Investigative Site, Pisa, PI, Italy
- Japan (12):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Sakaidechō, Kagawa-ken
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Habikino, Osaka
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- Netherlands (2):
  - Novartis Investigative Site, Harderwijk
  - Novartis Investigative Site, Leiden
- Slovakia (4):
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Liptovský Hrádok, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Zvolen

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to one of the four treatment arms.
Period: Overall Study
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Started | 2 | 2 | 3 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 3 | 3
Not completed — Study terminated. | 2 | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031 | Total
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.5 (16.26) | 47.0 (1.41) | 53.7 (11.59) | 47.7 (2.89) | 49.1 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 2 | 7
  Male | 0 | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: QGE031 Compared to Placebo in Atopic Asthma Patients on the Reduction in Rate of Severe Asthma Exacerbations
Time Frame: Week 52
Population: Due to the small number of patients randomized and limited treatment duration (not more than 22 days in QGE031 and 29 days in Placebo), the planned statistical analysis was not performed.
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: QGE031 Compared to Placebo in All Asthma Patients on the Reduction in Rate of Severe Asthma Exacerbations
Time Frame: Week 52
Population: as for outcome 1
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: QGE031 Compared to Placebo in Non-atopic Asthma Patients on the Reduction in Rate of Severe Asthma Exacerbations
Time Frame: Week 52
Population: as for outcome 1
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: QGE031 Compared to Placebo in Asthma Patients (All and Either Atopic or Non-atopic) on the Reduction in Rate of Asthma Exacerbations (by Severity)
Time Frame: Week 52
Population: as for outcome 1
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: QGE031 Compared to Placebo in Asthma Patients (All and Either Atopic or Non-atopic) on Time to First Asthma Exacerbations (by Severity)
Time Frame: Week 52
Population: as for outcome 1
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: QGE031 Compared to Placebo in Asthma Patients (All and Either Atopic or Non-atopic) on Change From Baseline in Asthma Control Questionnaire (ACQ)
Time Frame: Baseline, Treatment (Weeks 4, 8, 12, 16, 24, 36, 52), follow up (Weeks 60 and 72)
Population: as for outcome 1
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: QGE031 Compared to Placebo in Asthma Patients (All and Either Atopic or Non-atopic) on Change From Baseline in Asthma Control Diary (ACD)
Time Frame: Over 52 weeks (Treatment) and 20 weeks (follow-up)
Population: as for outcome 1
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: QGE031 Compared to Placebo in Asthma Patients (All and Either Atopic or Non-atopic) on Forced Expiratory Volume in 1 Second (FEV1)
Time Frame: Baseline, Treatment (Weeks 4, 8, 12, 16, 24, 36, 52), follow up (Weeks 60 and 72)
Population: as for outcome 1
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: QGE031 Compared to Placebo in Asthma Patients (All and Either Atopic or Non-atopic) on Peak Expiratory Flow (PEF) in the Morning and Evening
Time Frame: Over 52 weeks (Treatment) and 20 weeks (follow-up)
Population: as for outcome 1
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: QGE031 Compared to Placebo in Asthma Patients (All and Either Atopic or Non-atopic) on Total Daily Symptom Score
Time Frame: Over 52 weeks (Treatment) and 20 weeks (follow-up)
Population: as for outcome 1
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Response to QGE031 Between Atopic Asthma and Non-atopic Asthma
Time Frame: Over 52 weeks (treatment) and 20 weeks (follow up)
Population: as for outcome 1
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | QGE031 240 mg | QGE031 72 mg | QGE031 24 mg | Placebo to QGE031
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/2 | 2/2 | 1/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QGE031 240 mg (N=2) | QGE031 72 mg (N=2) | QGE031 24 mg (N=3) | Placebo to QGE031 (N=3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated due to the efficacy results from the Phase II study CQGE031B2201 (NCT01716754). Data analyses were not performed due to the very limited dataset (only 10 participants received study medication of the 440 participants planned).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.